CLINICAL TRIAL: NCT02830321
Title: Study to Explore the Association Between Hyperemesis Gravidarum in Pregnant Women and Helicobacter Pylori Infection by Using H.P. Stool Antigen Test to Diagnose H Pylori Infection
Brief Title: The Association of Helicobacter Pylori in the Pathogenesis of Hyperemesis Gravidarum in Pregnant Women
Acronym: AOHPIPOHGIPW
Status: Completed | Type: Observational
Sponsor: rasha fawzy abd el kader (Other)
Responsible Party: Sponsor-Investigator, rasha fawzy abd el kader, Principal Investigator, Ain Shams University
Organization: Ain Shams University (Other)
Other Study IDs: FDAAA
Record Dates: First submitted 2016-07-03; First posted 2016-07-12 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Hyperemesis Gravidarum
MeSH Terms: conditions — Hyperemesis Gravidarum

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- case: Pregnant women who suffered from hyperemesis gravidarum and admitted in the hospital
  * Age: 18-40 years old
  * Gestational age: less than 16 weeks confirmed by pelvic u/s
  * Excessive pregnancy - related nausea and /or vomiting that prevent adequate intake of food and fluids.
  All pregnant (case and control) were asked to bring a stool sample in a clean container. Collected samples were tested in a laboratory (Ain Shams Univerisity hospital).
  Stool samples were be tested by using one step H.pylori stool antigen test (CER TEST BIOTEC) for the detection of H. pylori antigen.
  Interventions: Other: helicopacter pylori stool antigen test (CER TEST BIOTEC)
- control: Control patients which are selected from pregnant women presenting to the outpatient clinics for routine antenatal care of the same gestational age, same age range and same socioeconomic standard as cases.
  Interventions: Other: helicopacter pylori stool antigen test (CER TEST BIOTEC)

INTERVENTIONS:
Other: helicopacter pylori stool antigen test (CER TEST BIOTEC) — Stool samples were tested by using one step H.pylori stool antigen test (CER TEST BIOTEC)for the detection of H. pylori antigen in pregnant women with hyperemesis gravidarum
  Other Names: (CER TEST BIOTEC)

SUMMARY:
The purpose of this study to explore the association between Hyperemesis Gravidarum in pregnant women and Helicobacter pylori infection.

DETAILED DESCRIPTION:
This study included 90 pregnant women during their first trimester who attended Ain Shams University Maternity Hospital antenatal clinic and admitted in the ward.

Patients were divided into two groups: 46 cases of pregnant women with H.G and 44 healthy control pregnant women with no vomiting.

Both groups were matched regarding the inclusion criteria which includes maternal age (18-40 years), gestational age (<16 wks), and signs and symptoms of H.G for cases (vomiting affecting the general condition, ketonuria, weight loss) and excluding cases or controls with multiple gestation, hyadatiform disease or maternal disease causes vomiting such as ; pyelonephritis, gastroenteritis, cholecystitis or hepatitis.

The two groups were subjected to full history taking, clinical examination, routine laboratory investigations (urine analysis, CBC, liver, kidney function tests Na, k, PT, PTT & INR) Abdominal ultrasound was done to assess fetal life and gestational age and to exclude gestational trophoblastic disease and multiple gestation pregnancy.H.Pylori infection was assessed by using One step H.pylori Stool Antigen Test.

(CER TEST BIOTEC) pol. Industrial Rio Gallego II,Calle J, No 1, 50840, San Mateo de Gallego, Zaragoza (SPAIN) for the detection of H. pylori antigen.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-40 years old
* Gestational age: less than 16 weeks confirmed by U/S
* Excessive pregnancy - related nausea and /or vomiting that prevent adequate intake of food and fluids.
* Measuring weight loss(>5% of pre-pregnancy weight)
* Signs of dehydration:

  * Ketonuria (+1 or more)
  * Hemoconcentration (normal Female hematocrit value (36.1-44.3%)

Exclusion Criteria:

* Multiple gestation pregnancy
* Hydatidiform molar pregnancy
* Other causes of vomiting:

  * Gastroentritis
  * Cholecystitis
  * Pyelonephritis
  * Liver dysfunction

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Study will include pregnant women in the first trimester attending Ain Shams University Maternity Hospital antenatal clinic and admitted in the ward.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2015-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The Association of Helicobacter Pylori in the Pathogenesis of Hyperemesis Gravidarum in Pregnant Women | from march 2015 to december 2015
  90 Participants were assessed by using H.p.S.Ag test to detect helicobacter infection in pregnant women

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Increased estrogen production causes decreased secretions of hydrochloric acids; therefore peptic ulcer formation or flare - up of existing peptic ulcers is uncommon during pregnancy and may improve (Winbery and Blaho, 2001).